CLINICAL TRIAL: NCT03861377
Title: "Hemodynamic Stability During Induction of General Anesthesia With Propofol and Remifentanil: A Randomized, Controlled, Double-blind Study Comparing Medium and Low Remifentanil Doses."
Brief Title: Hemodynamics During Induction of General Anesthesia With Medium or Low Remifentanil Doses.
Acronym: RH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helse Fonna (Other)
Responsible Party: Principal Investigator, Gunnar Helge Sjøen, Consultant in Anesthesiology, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2019/376; 2019-000961-19 (EudraCT Number)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Hemodynamic Instability; Anesthesia, General; Anesthesia, Intravenous
Keywords: Cardiac Output (CO); Systolic Blood Pressure (SBP); Systemic Vascular Resistance (SVR); Heart Rate (HR); Stroke Volume (SV); Lithium Dilutional Cardiac Output (LiDCO); Minimal Invasive Hemodynamic Monitor; Remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization made by a person not involved in trial in other ways. Allocation masked in sealed envelopes, stored in a locked cash box only opened by two drug preparing nurses not involved in patient care. Syringe labelled with patient identification (ID) (eg 03Remi). Patient, Care Provider and Investigator blinded for actual concentration of drug. Allocation break after data data wash and processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remifentanil R2 (Active Comparator): Low dose Remifentanil induction dose (R2)
  Interventions: Drug: Remifentanil R2
- Remifentanil R4 (Active Comparator): Medium dose Remifentanil induction dose (R4)
  Interventions: Drug: Remifentanil R4
- Remifentanil R8 (Active Comparator): Medium dose Remifentanil induction dose (R8)
  Interventions: Drug: Remifentanil R8

INTERVENTIONS:
Drug: Remifentanil R2 — 0,7 microg/kg
  Other Names: Ultiva
  Arms: Remifentanil R2
Drug: Remifentanil R4 — 1,1 microg/kg
  Other Names: Ultiva
  Arms: Remifentanil R4
Drug: Remifentanil R8 — 1,7 microg/kg
  Other Names: Ultiva
  Arms: Remifentanil R8

SUMMARY:
In this trial the investigators want to examine if there is any difference in hemodynamic stability during induction when comparing two low and a medium remifentanil dose and keeping propofol induction dose at about 2.0 mg/kg.

DETAILED DESCRIPTION:
Typically, one or more adjuvant medications is administered during induction of general anesthesia. When anesthetic drugs are combined, the hypnotic effects are often synergistic. Propofol is associated with hypotension and bradycardia and used together with remifentanil or sedative agents it may give synergistic or additive sedative and hemodynamic effects.

Remifentanil is infused at 0.05-0.3 microg/kg/min during induction of anesthesia. Some use a loading dose of 0.5-1.0 microg/kg before starting the continuous infusion. The onset of action of remifentanil is within one to two minutes and it reaches rapidly a steady state effect site concentration after a bolus dose.

Kazmaier (2000) showed that a high-dose remifentanil anesthesia (2 microg/kg/min) reduced cardiac index (-25%), stroke volume (-14%) and mean arterial blood pressure (-39%) in a similar manner as propofol/remifentanil (propofol target 2 microg/ml and remifentanil 0.5 microg/kg/min), but systemic vascular resistance index decreased (-14%) in propofol/remifentanil combination. Fairfield et al have earlier (1991) showed that propofol 2.5 mg/kg induction without opioid reduces cardiac output (-15%) stroke volume (-5 %), mean arterial pressure (-33%) and systemic vascular resistance (-11%) and a slight reduction i heart rate. Guarracino (2003) suggests the reduction in cardiac index during induction with propofol/remifentanil with a low propofol target (1.2 microg/ml) may be due to decreased heart rate. Zaballos (2009) have shown that remifentanil depresses sinus node and atrioventricular (AV) -nodal function in comparison with propofol alone in a closed chest porcine model. Hayashi (2016) states that even in a low remifentanil effect site concentration (3.5 nanog/ml) it may reduce heart rate significantly when combined with propofol bolus 30-50 mg.

ELIGIBILITY:
Inclusion Criteria:

* Gynecological procedure
* Age 18-50 years
* General anesthesia planned
* Systolic blood pressure < 150 mmHg, HR < 100 beats/min

Exclusion Criteria:

* Pre-existing hypertension
* Diabetes
* Ischemic heart disease or cerebrovascular disease
* Heart valve disease
* Verified cardiac arrhythmia other than extrasystoles
* Verified anaemia with hemoglobin level below 9.0 gr/dl.
* Kidney or hepatic disease
* Hypersensitivity for propofol, soya, eggs or peanuts
* Pregnancy
* Poor health state
* Illicit substance use
* BMI <20 or >35 kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) | First 7,5 minutes from start of induction
  Change in systolic blood pressure during induction
Heart Rate (HR) | First 7,5 minutes from start of induction
  Change in heart rate during induction

SECONDARY OUTCOMES:
Stroke Volume (SV) | First 7,5 minutes from start of induction
  Change in stroke volume during induction
Cardiac Output (CO) | First 7,5 minutes from a start of induction
  Change in cardiac output during induction
Systemic Vascular Resistance (SVR) | First 7,5 minutes from start of induction
  Change in systemic vascular resistance during induction

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Sjøen, MD, Principal Investigator — Helse Fonna
Locations (1):
- Kirurgisk Klinikk Anestesi, Haugesund, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
LiDCO-csv raw data and processed data will be made public at the publishers site, and the supporting information by request to the Principal Investigator. Statistical Data Plan is included in Study Protocol.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be stored for 15 years after end of study, and may be shared during this time frame.
Access Criteria: The data may be shared by contacting the Principal Investigator.

REFERENCES:
- [Background] Kazmaier S, Hanekop GG, Buhre W, Weyland A, Busch T, Radke OC, Zoelffel R, Sonntag H. Myocardial consequences of remifentanil in patients with coronary artery disease. Br J Anaesth. 2000 May;84(5):578-83. doi: 10.1093/bja/84.5.578. PMID 10844832
- [Background] Fairfield JE, Dritsas A, Beale RJ. Haemodynamic effects of propofol: induction with 2.5 mg kg-1. Br J Anaesth. 1991 Nov;67(5):618-20. doi: 10.1093/bja/67.5.618. PMID 1751277
- [Background] Guarracino F, Penzo D, De Cosmo D, Vardanega A, De Stefani R. Pharmacokinetic-based total intravenous anaesthesia using remifentanil and propofol for surgical myocardial revascularization. Eur J Anaesthesiol. 2003 May;20(5):385-90. doi: 10.1017/s0265021503000589. PMID 12790210
- [Background] Zaballos M, Jimeno C, Almendral J, Atienza F, Patino D, Valdes E, Navia J, Anadon MJ. Cardiac electrophysiological effects of remifentanil: study in a closed-chest porcine model. Br J Anaesth. 2009 Aug;103(2):191-8. doi: 10.1093/bja/aep131. Epub 2009 May 20. PMID 19457895
- [Background] Hayashi K, Tanaka A. Effect-site concentrations of remifentanil causing bradycardia in hypnotic and non-hypnotic patients. J Clin Monit Comput. 2016 Dec;30(6):919-924. doi: 10.1007/s10877-015-9794-4. Epub 2015 Oct 13. PMID 26462495